CLINICAL TRIAL: NCT00720954
Title: Rigid Thoracoscopy Versus CT-Guided Pleural Needle Biopsy For Diagnosis of Patients With Pleural Effusions: A Randomized Control Trial
Brief Title: Rigid Thoracoscopy Versus CT-Guided Pleural Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Dr. Muzaffer Metintas
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: 2007.11.008
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Pleural Effusion; Pleural Diseases
Keywords: Thoracoscopy; Pleural needle biopsy; Malignant pleural diseases; Mesothelioma; Diagnosis; Pleurisy tuberculosis; Patients with pleural diseases and pleural effusion should have been included in the study.
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases; Mesothelioma; Disease | interventions — Clinical Laboratory Techniques; Thoracoscopy

ARMS (2):
- A (Other): CT guided pleural needle biopsy
  Interventions: Procedure: Ct-guided pleural needle biopsy
- B (Other): Thoracoscopy
  Interventions: Procedure: Thoracoscopy

INTERVENTIONS:
Procedure: Ct-guided pleural needle biopsy — Biopsy of pleura
  Other Names: Diagnose
  Arms: A
Procedure: Thoracoscopy — Biopsy of pleura
  Other Names: Diagnose
  Arms: B

SUMMARY:
The aim of this study is to compare the rigid thoracoscopy with CT-guided pleural needle biopsy by the diagnostic efficacy and safety in patients with pleural effusion.

DETAILED DESCRIPTION:
Pleural needle biopsy with Abrams needle, which can be performed by all chest physicians, is a simple, safe and cheap method of obtaining tissue from pleura, but its diagnostic rate is between 7 % -72 %, ~ 50 %. Problems for Abrams needle are scattered tumoral involvement on pleura, blind performance, small tissue sampling, to tend to early and dense fibrosis and usually involvement of lower pleural surface and diaphragmatic pleura.

Pleural needle biopsy with Abrams' needle, which can be performed by all chest physicians, if done with image guided and if this increase the diagnosis rate, the number of second procedure which is more expensive and hard will decrease.

The study aims the comparison of rigid thoracoscopy with CT-guided pleural needle biopsy by the diagnostic efficacy and safety in patients with pleural effusion.

It has been planned that a total of 120 patients accepted to the study who have pleural effusion at plain chest roentgenogram. All patients are being randomized after underwent contrast-enhanced CT. Undiagnosed patients of biopsy group are performed thoracoscopy and undiagnosed patients of thoracoscopy group followed up.

Two groups will compare by age, sex, Karnofsky performance status (KPS), diagnosis and complication rate.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18-85
2. Pleural effusion in conventional radiography
3. At least 10x10 cm space in pleural space with effusion
4. No bleeding diathesis
5. Informed consent

Exclusion Criteria:

1. Patients who went under pleural biopsy before
2. Arrythmia
3. Hypertensive attack during biopsy
4. Bleeding diathesis
5. Hypoxemia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of both thoracoscopy and CT-guided pleural needle biopsy for diagnosis of pleural diseases | 30 months

SECONDARY OUTCOMES:
Determine the efficacy of pleural needle biopsy and thoracoscopy in relation to CT findings. | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- ESOGU MEDICAL FACULTY DEPARTMENT of CHEST DISEASES, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Derived] Metintas M, Ak G, Dundar E, Yildirim H, Ozkan R, Kurt E, Erginel S, Alatas F, Metintas S. Medical thoracoscopy vs CT scan-guided Abrams pleural needle biopsy for diagnosis of patients with pleural effusions: a randomized, controlled trial. Chest. 2010 Jun;137(6):1362-8. doi: 10.1378/chest.09-0884. Epub 2010 Feb 12. PMID 20154079
- See also: University — http://www.ogu.edu.tr